CLINICAL TRIAL: NCT01643772
Title: OxyNorm® Capsules (Immediate-Release) PK Study
Brief Title: OxyNorm® Capsules (Immediate-Release) Pharmacokinetic (PK) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXYC09-CN-102
Record Dates: First submitted 2011-11-17; First posted 2012-07-18 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxycodone Hydrochloride 5 mg Capsules (Experimental): Group 1: single dose Oxycodone Hydrochloride 5 mg Capsules after 10 hours fasting
  Interventions: Drug: Oxycodone hydrochloride
- Oxycodone Hydrochloride 10 mg Capsules (Experimental): Group 2: single dose Oxycodone Hydrochloride 10 mg Capsules after 10 hours fasting
  Interventions: Drug: Oxycodone hydrochloride
- Oxycodone Hydrochloride 20 mg Capsules (Experimental): Group 3: single dose Oxycodone Hydrochloride 20 mg Capsules after 10 hours fasting
  Interventions: Drug: Oxycodone hydrochloride
- Oxycodone Hydrochloride 10 mg Capsules(multi-dose) (Experimental): Group 4: multi-dose 4 times per day Oxycodone Hydrochloride 10mg Capsules for 3 days, and one dose on 4th day morning
  Interventions: Drug: Oxycodone hydrochloride

INTERVENTIONS:
Drug: Oxycodone hydrochloride — The subjects will be randomized to receive either a single dose of OxyNorm® Capsules 5, 10, 20mg, or multiple-dose OxyNorm® Capsules 10 mg for 13 times.
  Other Names: OxyNorm® Capsules

SUMMARY:
A Single Dose PK Study of OxyNorm® immediate-release capsules 5, 10, and 20mg, and a multiple-dose PK Study of OxyNorm® immediate-release capsules 10mg in Chinese patients with pain.It will be a single center, open label, randomized, oral administration study.

DETAILED DESCRIPTION:
Single dose: The subjects will be randomized to receive a single dose of OxyNorm® immediate-release capsules 5, 10, and 20mg.

Multiple dose: The subjects will take 3 days OxyNorm® capsule 10mg, once every 6 hours, 10mg per dose. In the morning of the 4th day, the subjects will take single dose of OxyNorm® capsule 10mg. On the 5th day, all the subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain, Multiple dose group should enroll the Patients with cancer pain;
* Patients aged >≥30 to ≤ 60 years;
* Body weight ≥ 45kg, and BMI range ≥19, <24;
* Karnofsky score ≥ 70;
* The results of liver function and kidney tests must meet the following criteria: ALT、AST is within the upper limit of normal value ranges by a factor 2, and TB、BUN、Cr is within the upper limit of normal value ranges by a factor 1.25;
* The electrocardiogram examination results are normal;
* Patients must have given a written informed consent prior to this trial, and have the capability to complete every required test.

Exclusion Criteria:

* Have hypersensitivity history to any opioids;
* Have known hypersensitivity to any of compositions of the study drugs;
* Patients who are likely to have paralytic ileus or acute abdomen or to perform an operation on abdominal region；
* Patients with respiratory depression, cor pulmonale, or chronic bronchial asthma;
* Patients who are unable to stop taking monoamine oxidase inhibitor during this trial period or time lapses less than 2 weeks since drug withdrawal;
* Patients with hypercarbia;
* Patients with biliary tract diseases, pancreatitis, prostatic hypertrophy, or corticoadrenal insufficiency;
* Patients with alcoholism or drug abuse history;
* Positive anti-HIV or syphilis antibody test result;
* Patients who are pregnant, or lactating;
* Urine screening before study is positive for opioids, barbiturates, amphetamines, cocaine metabolites, methadone, diazepam and cannabinoids;
* Donated 400 mL or more of blood or blood products within 3 months prior to the start of the study, or donated 200 mL or more of blood or blood products within one month prior to the start of the study;
* Subjects who participated in a clinical research study within one month of study entry;
* Patients who are currently taking opioids.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mundipharma China Ltd., Study Chair — Mundipharma China Ltd.
Locations (1):
- Affiliated Hospital to Academy of Military Medical Science of China People's Liberation Army, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in phase I unit in two public hospitals, the first subject took the first dose study medication on 13May2011, the last subject took the last dose on 6Jul2012.
Pre-assignment Details: The study has a 7-days screening phase, for the subject who meet all the inclusion and exclusion criteria was dosed without run-in or wash out period.
Groups:
- Oxycodone Hydrochloride Single Dose(5mg): Group 1: single dose Oxycodone Hydrochloride 5 mg Capsules after 10 hours fasting
- Oxycodone Hydrochloride Single Dose(10mg): Group 2: single dose Oxycodone Hydrochloride 10 mg Capsules after 10 hours fasting
- Oxycodone Hydrochloride Single Dose(20mg): Group 3: single dose Oxycodone Hydrochloride 20 mg Capsules after 10 hours fasting
- Oxycodone Hydrochloride Multiple Dose: Group 4: multi-dose 4 times per day Oxycodone Hydrochloride 10mg Capsules for 3 days, and one dose on 4th day morning
Period: Overall Study
Arm/Group | Oxycodone Hydrochloride Single Dose(5mg) | Oxycodone Hydrochloride Single Dose(10mg) | Oxycodone Hydrochloride Single Dose(20mg) | Oxycodone Hydrochloride Multiple Dose
Started | 15 | 15 | 15 | 16
Completed | 15 | 15 | 15 | 14
Not Completed | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: PP Population
Groups:
- Oxycodone Hydrochloride Multiple Dose(10mg): Group 4: multi-dose 4 times per day Oxycodone Hydrochloride 10mg Capsules for 3 days, and one dose on 4th day morning
- Total: Total of all reporting groups
Arm/Group | Oxycodone Hydrochloride Single Dose(5mg) | Oxycodone Hydrochloride Single Dose(10mg) | Oxycodone Hydrochloride Single Dose(20mg) | Oxycodone Hydrochloride Multiple Dose(10mg) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 61
Age, Continuous [Mean (Standard Deviation); unit: year] — Population: PP population
  year
    number analyzed (Participants) | 15 | 15 | 14 | 14 | 58
    (all) | 40.22 (4.90) | 39.63 (6.21) | 36.16 (8.68) | 48.62 (7.87) | 41.11 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: PP Population
  Participants
    number analyzed (Participants) | 15 | 15 | 14 | 14 | 58
    Female | 8 | 8 | 5 | 7 | 28
    Male | 7 | 7 | 9 | 7 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: PP Population
  Participants
    number analyzed (Participants) | 15 | 15 | 14 | 14 | 58
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 15 | 15 | 14 | 14 | 58
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: PP Population
  participants
    China: number analyzed (Participants) | 15 | 15 | 14 | 14 | 58
    China | 15 | 15 | 14 | 14 | 61

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t and AUC0-∞ for Participants Who Received a Single Dose
Description: To calculate AUC0-t AUC0-∞of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method.Plasma concentrations of Oxycodone Hydrochloride single dose 5mg,10mg,20mg will be analyzed.
Time Frame: blood sample at predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24hr post-dose.
Population: PP Population
Measure: Mean (Standard Deviation); unit: ng*hr*ml
Groups:
- Oxycodone Hydrochloride Single Dose 5 mg: Group 1: single dose Oxycodone Hydrochloride 5 mg Capsules after 10 hours fasting
- Oxycodone Hydrochloride Single Dose 10 mg: Group 2: single dose Oxycodone Hydrochloride 10 mg Capsules after 10 hours fasting
- Oxycodone Hydrochloride Single Dose 20 mg: Group 3: single dose Oxycodone Hydrochloride 20 mg Capsules after 10 hours fasting
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
ng*hr*ml
  Oxycondone(AUC0-t) | 57.03 (14.62) | 102.10 (23.94) | 205.89 (58.03)
  Oxycondone(AUC0-∞) | 58.38 (15.41) | 104.56 (25.16) | 210.61 (59.89)
  Noroxycodone(AUC0-t): number analyzed (Participants) | 14 | 15 | 14
  Noroxycodone(AUC0-t) | 38.85 (9.61) | 89.76 (29.13) | 163.68 (43.29)
  Noroxycodone(AUC0-∞) | 41.93 (11.09) | 99.15 (34.11) | 178.61 (46.70)
  Hydroxymorphine(AUC0-t): number analyzed (Participants) | 0 | 1 | 1
  Hydroxymorphine(AUC0-t) |  | 3.12 (0) | 3.79 (0)
  Hydroxymorphine(AUC0-∞) | 0 (0) | 3.96 (0) | 4.36 (0)
  Normethoxymorphone(AUC0-t): number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone(AUC0-t) | 13.27 (10.43) | 28.69 (26.39) | 37.64 (17.51)
  Normethoxymorphone(AUC0-∞): number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone(AUC0-∞) | 15.07 (11.54) | 33.31 (29.29) | 43.85 (19.42)

2. Primary Outcome: Cmax,Clast for Participants Who Received a Single Dose
Description: To calculate Cmax,Clast of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in single dose 5mg,10mg,20mg.
Time Frame: blood sample at predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24hr post-dose.
Population: PP population
Measure: Mean (Standard Deviation); unit: ng*mL
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
ng*mL
  Oxycodone(Cmax) | 12.97 (2.67) | 21.14 (4.58) | 35.56 (14.18)
  Noroxycodone(Cmax) | 6.19 (2.15) | 11.62 (2.79) | 19.19 (5.88)
  Hydroxymorphine(Cmax) | 0.27 (0.12) | 0.42 (0.20) | 0.76 (0.29)
  Normethoxymorphone(Cmax) | 1.64 (1.52) | 1.77 (1.46) | 3.52 (1.75)
  Oxycodone(Clast) | 0.20 (0.11) | 0.37 (0.20) | 0.74 (0.30)
  Noroxycodone(Clast) | 0.32 (0.17) | 0.89 (0.51) | 1.56 (0.47)
  Hydroxymorphine(Clast): number analyzed (Participants) | 0 | 1 | 1
  Hydroxymorphine(Clast) |  | 0.05 (0) | 0.05 (0)
  Normethoxymorphone(Clast): number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone(Clast) | 0.16 (0.12) | 0.36 (0.28) | 0.49 (0.25)

3. Primary Outcome: Tmax,t1/2 for Participants Who Received a Single Dose
Description: To calculate Tmax,t1/2 of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in single dose 5mg,10mg,20mg.
Time Frame: blood sample at predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24hr post-dose.
Population: PP popluation
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
hour
  Oxycodone (Tmax) | 0.98 (0.43) | 0.80 (0.22) | 0.73 (0.18)
  Oxycodone (t1/2) | 4.42 (0.70) | 4.38 (0.57) | 4.24 (0.52)
  Noroxycodone (Tmax) | 1.32 (1.36) | 1.08 (0.82) | 0.98 (0.64)
  Noroxycodone (t1/2) | 6.22 (1.18) | 6.63 (1.47) | 6.59 (0.61)
  Hydroxymorphine(Tmax) | 0.90 (0.32) | 0.87 (0.33) | 1.07 (0.94)
  Hydroxymorphine (t1/2): number analyzed (Participants) | 0 | 1 | 1
  Hydroxymorphine (t1/2) |  | 11.70 (0) | 7.90 (0)
  Normethoxymorphone(Tmax) | 1.62 (1.38) | 1.77 (1.46) | 2.04 (1.84)
  Normethoxymorphone(t1/2): number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone(t1/2) | 7.78 (1.71) | 9.17 (1.93) | 8.22 (2.28)

4. Primary Outcome: Clearance Rate for Participants Who Received a Single Dose
Description: To calculate CL of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in single dose 5mg,10mg,20mg.
Time Frame: blood sample at predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24hr post-dose.
Population: PP popuplation
Measure: Mean (Standard Deviation); unit: L*hour
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
L*hour
  Oxycodone (CL) | 91.49 (24.45) | 101.53 (27.54) | 101.33 (25.16)
  Noroxycodone (CL) | 125.78 (28.40) | 113.30 (40.85) | 119.38 (31.09)
  Hydroxymorphine(CL): number analyzed (Participants) | 0 | 1 | 1
  Hydroxymorphine(CL) |  | 2525.30 (0) | 4587.50 (0)
  Normethoxymorphone(CL): number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone(CL) | 443.45 (192.68) | 530.65 (368.02) | 681.64 (736.51)

5. Primary Outcome: Vd for Participants Who Received a Single Dose
Description: To calculate Apparent Distribution Volume (Vd) Vd of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in single dose 5mg,10mg,20mg.
Time Frame: blood sample at predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24hr post-dose.
Population: PP population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
L
  Oxycodone | 568.11 (118.51) | 626.45 (115.70) | 611.17 (137.94)
  Noroxycodone | 1119.22 (312.37) | 1026.65 (230.16) | 1138.72 (335.51)
  Hydroxymorphine: number analyzed (Participants) | 0 | 1 | 1
  Hydroxymorphine |  | 42608.80 (0) | 52264.20 (0)
  Normethoxymorphone: number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone | 5004.50 (2443.16) | 7297.56 (5341.91) | 7460.04 (5956.86)

6. Primary Outcome: ke for Participants Who Received a Single Dose
Description: To calculate Terminal Elimination Rate (ke) of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in single dose 5mg,10mg,20mg.
Time Frame: blood sample at predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24hr post-dose.
Population: PP population
Measure: Mean (Standard Deviation); unit: h^-1
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
h^-1
  Oxycodone | 0.16 (0.03) | 0.16 (0.02) | 0.17 (0.02)
  Noroxycodone | 0.12 (0.02) | 0.11 (0.02) | 0.11 (0.01)
  Hydroxymorphine: number analyzed (Participants) | 0 | 1 | 1
  Hydroxymorphine |  | 0.06 (0) | 0.09 (0)
  Normethoxymorphone: number analyzed (Participants) | 14 | 14 | 14
  Normethoxymorphone | 0.09 (0.02) | 0.08 (0.02) | 0.10 (0.05)

7. Primary Outcome: AUCss for Participants Who Received Multiple Dose
Description: To calculate AUCss of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in multiple dose 10mg.
Time Frame: Predose for the 1st, 2nd, 3rd day and predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24 post dose on the 4th day.
Population: PP population
Measure: Mean (Standard Deviation); unit: ng*hours*mL
Arm/Group | Oxycodone Hydrochloride Multiple Dose
Number analyzed (Participants) | 14
ng*hours*mL
  Oxycodone | 156.03 (72.07)
  Noroxycodone | 122.69 (39.02)
  Hydroxymorphine: number analyzed (Participants) | 7
  Hydroxymorphine | 4.51 (1.40)
  Normethoxymorphone | 16.56 (8.34)

8. Primary Outcome: Css_min,Css_max and Css_av for Participants Who Received Multiple Dose
Description: To calculate Css_min,Css_max and Css_av of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in multiple dose 10mg.
Time Frame: Predose for the 1st, 2nd, 3rd day and predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24 post dose on the 4th day.
Population: multiple dose group has 14 subjects
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Oxycodone Hydrochloride Multiple Dose
Number analyzed (Participants) | 14
ng/ml
  Oxycodone(Css_min) | 16.92 (8.71)
  Noroxycodone(Css_min) | 15.74 (5.58)
  Hydroxymorphine(Css_min): number analyzed (Participants) | 7
  Hydroxymorphine(Css_min) | 0.40 (0.20)
  Normethoxymorphone(Css_min) | 2.18 (1.02)
  Oxycodone(Css_max ) | 40.17 (15.38)
  Noroxycodone(Css_max ) | 26.71 (8.03)
  Hydroxymorphine(Css_max ) | 1.10 (0.47)
  Normethoxymorphone(Css_max ) | 3.65 (1.97)
  Oxycodone(Css_av) | 26.01 (12.01)
  Noroxycodone(Css_av) | 20.44 (6.50)
  Hydroxymorphine(Css_av) | 0.75 (0.24)
  Normethoxymorphone(Css_av) | 2.76 (1.39)

9. Primary Outcome: Tmax,t1/2 for Participants Who Received Multiple Dose
Description: To calculate Tmax,t1/2 of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in multiple dose 10mg.
Time Frame: Predose for the 1st, 2nd, 3rd day and predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24 post dose on the 4th day.
Population: multiple dose group has 14 subjects
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Oxycodone Hydrochloride Multiple Dose
Number analyzed (Participants) | 14
hour
  Oxycodone( Tmax) | 1.35 (0.65)
  Noroxycodone( Tmax) | 1.51 (1.00)
  Hydroxymorphine( Tmax) | 1.49 (1.00)
  Normethoxymorphone( Tmax) | 1.86 (1.48)
  Oxycodone(t1/2) | 5.07 (1.47)
  Noroxycodone(t1/2) | 7.23 (1.92)
  Hydroxymorphine(t1/2) | 8.09 (2.60)
  Normethoxymorphone(t1/2) | 9.07 (1.96)

10. Primary Outcome: CL for Participants Who Received Multiple Dose
Description: To calculate Clearance rate (CL) of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in multiple dose 10mg.
Time Frame: Predose for the 1st, 2nd, 3rd day and predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24 post dose on the 4th day.
Population: multiple dose group has 14 subjects
Measure: Mean (Standard Deviation); unit: L*hour
Arm/Group | Oxycodone Hydrochloride Multiple Dose
Number analyzed (Participants) | 14
L*hour
  Oxycodone | 73.54 (24.08)
  Noroxycodone | 90.66 (32.56)
  Hydroxymorphine: number analyzed (Participants) | 7
  Hydroxymorphine | 2374.20 (597.75)
  Normethoxymorphone | 773.01 (431.19)

11. Primary Outcome: Fluctuation Index (DF) for Participants Who Received Multiple Dose
Description: To calculate Fluctuation index (DF) of Drug Valley and Peak Concentration of Oxycondone,Noroxycodone,Hydroxymorphine, Normethoxymorphone with Non-atrioventricular model method in multiple dose 10mg.
Time Frame: Predose for the 1st, 2nd, 3rd day and predose,15min,30min,45min,1,1.5,2,3,4,6,8,12,24 post dose on the 4th day.
Population: multiple dose group has 14 subjects
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Oxycodone Hydrochloride Multiple Dose
Number analyzed (Participants) | 14
ng/ml
  Oxycodone | 94.11 (32.64)
  Noroxycodone | 55.75 (23.54)
  Hydroxymorphine: number analyzed (Participants) | 7
  Hydroxymorphine | 123.95 (57.22)
  Normethoxymorphone | 52.07 (37.68)

12. Primary Outcome: The Excretion of Oxycondone, Noroxycodone, Hydroxymorphine,Normethoxymorphone in Urine(Single Dose)
Description: The excretion of drugs were calculated according to the concentration and volume of drugs in urine after single dose.
Time Frame: Pre-dose,post dose0-2h,post dose2-4h,post dose4-8h,post dose8-12h,post dose12-24h
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
μg
  Oxycondone(Pre-dose) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Oxycondone(post dose0-2h) | 25.69 (29.55) | 54.55 (79.39) | 108.57 (171.53)
  Oxycondone(post dose2-4h) | 64.24 (72.40) | 172.38 (192.35) | 316.07 (188.88)
  Oxycondone(post dose4-8h) | 64.93 (56.60) | 169.28 (268.13) | 165.45 (101.00)
  Oxycondone(post dose8-12h) | 56.07 (84.81) | 78.48 (91.91) | 71.07 (76.02)
  Oxycondone(post dose12-24h) | 40.30 (88.58) | 36.12 (33.66) | 67.92 (86.71)
  Noroxycodone(Pre-dose) | 0 (0) | 0 (0) | 0 (0)
  Noroxycodone(post dose0-2h) | 23.29 (39.94) | 63.80 (83.33) | 157.75 (229.32)
  Noroxycodone(post dose2-4h) | 105.53 (112.06) | 346.22 (262.65) | 784.70 (390.56)
  Noroxycodone(post dose4-8h) | 153.49 (124.65) | 418.95 (527.24) | 712.81 (417.09)
  Noroxycodone(post dose8-12h) | 139.45 (138.45) | 212.68 (170.80) | 360.37 (375.81)
  Noroxycodone(post dose12-24h) | 53.09 (41.21) | 128.75 (90.37) | 265.31 (400.05)
  Hydroxymorphine(Pre-dose) | 0 (0) | 0 (0) | 0 (0)
  Hydroxymorphine(post dose0-2h) | 0.51 (0.65) | 0.94 (1.41) | 2.89 (4.87)
  Hydroxymorphine(post dose2-4h) | 1.03 (1.03) | 2.52 (3.02) | 9.99 (7.14)
  Hydroxymorphine(post dose4-8h) | 1.72 (1.46) | 5.80 (12.62) | 5.85 (6.09)
  Hydroxymorphine(post dose8-12h) | 2.07 (3.39) | 2.97 (4.02) | 2.49 (2.62)
  Hydroxymorphine(post dose12-24h) | 2.31 (6.15) | 1.67 (1.86) | 2.90 (3.74)
  Normethoxymorphone(Pre-dose) | 0 (0) | 0 (0) | 0 (0)
  Normethoxymorphone(post dose0-2h) | 3.97 (6.96) | 7.16 (11.48) | 8.53 (13.63)
  Normethoxymorphone(post dose2-4h) | 15.44 (12.78) | 23.53 (16.86) | 40.29 (33.67)
  Normethoxymorphone(post dose4-8h) | 25.15 (33.82) | 68.87 (131.24) | 39.64 (23.90)
  Normethoxymorphone(post dose8-12h) | 28.59 (30.00) | 30.17 (21.62) | 48.38 (49.36)
  Normethoxymorphone(post dose12-24h) | 26.74 (30.33) | 30.16 (34.28) | 33.76 (31.67)

13. Primary Outcome: Cumulative Excretion of Oxycondone, Noroxycodone, Hydroxymorphine,Normethoxymorphone in Urine(Single Dose)
Description: Cumulative excretion of drugs were calculated according to the concentration and volume of drugs in urine after single dose.
Time Frame: post dose0-2h,post dose2-4h,post dose4-8h,post dose8-12h,post dose12-24h
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
μg
  Oxycondone(post dose0-2h) | 25.69 (29.55) | 54.55 (79.39) | 108.57 (171.53)
  Oxycondone(post dose2-4h) | 89.93 (91.36) | 226.92 (244.12) | 424.64 (326.09)
  Oxycondone(post dose4-8h) | 154.86 (129.52) | 396.20 (410.41) | 590.08 (361.27)
  Oxycondone(post dose8-12h) | 210.92 (203.25) | 474.68 (455.83) | 661.15 (338.34)
  Oxycondone(post dose12-24h) | 251.22 (198.78) | 510.80 (462.41) | 729.07 (343.84)
  Noroxycodone(post dose0-2h) | 23.29 (39.94) | 63.80 (83.33) | 157.75 (229.32)
  Noroxycodone(post dose2-4h) | 128.82 (117.04) | 410.02 (283.62) | 942.44 (529.85)
  Noroxycodone(post dose4-8h) | 282.31 (192.38) | 828.97 (629.00) | 1655.25 (736.42)
  Noroxycodone(post dose8-12h) | 421.75 (222.63) | 1041.66 (699.41) | 2015.62 (865.69)
  Noroxycodone(post dose12-24h) | 474.85 (232.06) | 1170.41 (703.51) | 2280.92 (936.47)
  Hydroxymorphine(post dose0-2h) | 0.51 (0.65) | 0.94 (1.41) | 2.89 (4.87)
  Hydroxymorphine(post dose2-4h) | 1.54 (1.56) | 3.46 (3.79) | 12.88 (10.40)
  Hydroxymorphine(post dose4-8h) | 3.27 (2.47) | 9.27 (13.89) | 18.73 (15.23)
  Hydroxymorphine(post dose8-12h) | 5.33 (4.83) | 12.24 (16.33) | 21.22 (15.56)
  Hydroxymorphine(post dose12-24h) | 7.64 (6.81) | 13.91 (17.13) | 24.11 (15.73)
  Normethoxymorphone(post dose0-2h) | 3.97 (6.96) | 7.16 (11.48) | 8.53 (13.63)
  Normethoxymorphone(post dose2-4h) | 19.40 (18.45) | 30.68 (19.15) | 48.82 (40.37)
  Normethoxymorphone(post dose4-8h) | 44.55 (44.62) | 99.55 (143.15) | 88.46 (53.96)
  Normethoxymorphone(post dose8-12h) | 73.14 (58.19) | 129.72 (154.63) | 136.84 (65.32)
  Normethoxymorphone(post dose12-24h) | 99.87 (76.02) | 159.88 (184.11) | 170.60 (74.03)

14. Primary Outcome: Average Cumulative Excretion Rate of Oxycondone, Noroxycodone, Hydroxymorphine,Normethoxymorphone in Urine(Single Dose)
Description: Average cumulative excretion rate of drugs were calculated according to the concentration and volume of drugs in urine after single dose.
Time Frame: post dose 24h
Measure: Mean (Standard Deviation); unit: % of ug
Arm/Group | Oxycodone Hydrochloride Single Dose 5 mg | Oxycodone Hydrochloride Single Dose 10 mg | Oxycodone Hydrochloride Single Dose 20 mg
Number analyzed (Participants) | 15 | 15 | 14
% of ug
  Oxycondone | 5.02 (3.98) | 5.11 (4.62) | 3.65 (1.72)
  Noroxycodone | 9.50 (4.64) | 11.70 (7.04) | 11.40 (4.68)
  Hydroxymorphine | 0.15 (0.14) | 0.14 (0.17) | 0.12 (0.08)
  Normethoxymorphone | 2.00 (1.52) | 1.60 (1.84) | 0.85 (0.37)

15. Primary Outcome: The Excretion of Oxycondone, Noroxycodone, Hydroxymorphine,Normethoxymorphone in Urine(Multiple Dose)
Description: The excretion of drugs were calculated according to the concentration and volume of drugs in urine after multiple dose on the 4th day.
Time Frame: Pre-dose,post dose0-2h,post dose2-4h,post dose4-8h,post dose8-12h,post dose12-24h on the 4th day
Measure: Mean (Standard Deviation); unit: μg
Groups:
- Oxycodone Hydrochloride Multiple Dose 10 mg: Group 2: multiple dose Oxycodone Hydrochloride 10 mg Capsules after 10 hours fasting
Arm/Group | Oxycodone Hydrochloride Multiple Dose 10 mg
Number analyzed (Participants) | 14
μg
  Oxycondone(Pre-dose) | 745.99 (1106.32)
  Oxycondone(post dose0-2h) | 263.32 (236.25)
  Oxycondone(post dose2-4h) | 342.64 (301.21)
  Oxycondone(post dose4-8h) | 431.70 (532.48)
  Oxycondone(post dose8-12h) | 137.13 (107.95)
  Oxycondone(post dose12-24h) | 344.15 (516.94)
  Noroxycodone(Pre-dose) | 897.44 (1121.80)
  Noroxycodone(post dose0-2h) | 372.51 (290.26)
  Noroxycodone(post dose2-4h) | 438.24 (218.90)
  Noroxycodone(post dose4-8h) | 515.39 (423.80)
  Noroxycodone(post dose8-12h) | 500.42 (717.43)
  Noroxycodone(post dose12-24h) | 865.37 (861.94)
  Hydroxymorphine(Pre-dose) | 9.43 (10.39)
  Hydroxymorphine(post dose0-2h) | 6.13 (8.11)
  Hydroxymorphine(post dose2-4h) | 24.03 (59.61)
  Hydroxymorphine(post dose4-8h) | 24.52 (27.45)
  Hydroxymorphine(post dose8-12h) | 15.10 (17.60)
  Hydroxymorphine(post dose12-24h) | 31.73 (36.65)
  Normethoxymorphone(Pre-dose) | 337.01 (460.24)
  Normethoxymorphone(post dose0-2h) | 130.63 (100.61)
  Normethoxymorphone(post dose2-4h) | 208.27 (183.64)
  Normethoxymorphone(post dose4-8h) | 262.56 (382.79)
  Normethoxymorphone(post dose8-12h) | 102.36 (91.74)
  Normethoxymorphone(post dose12-24h) | 240.75 (332.72)

16. Primary Outcome: Cumulative Excretion of Oxycondone, Noroxycodone, Hydroxymorphine,Normethoxymorphone in Urine(Mutilple Dose)
Description: Cumulative excretion of drugs were calculated according to the concentration and volume of drugs in urine after multiple dose on the 4th day .
Time Frame: post dose0-2h,post dose2-4h,post dose4-8h,post dose8-12h,post dose12-24h on the 4th day
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Oxycodone Hydrochloride Single Dose 10 mg
Number analyzed (Participants) | 14
μg
  Oxycondone(post dose0-2h) | 263.32 (236.25)
  Oxycondone(post dose2-4h) | 605.96 (479.83)
  Oxycondone(post dose4-8h) | 1037.66 (985.45)
  Oxycondone(post dose8-12h) | 913.59 (374.77)
  Oxycondone(post dose12-24h) | 1290.63 (720.65)
  Noroxycodone(post dose0-2h) | 372.51 (290.26)
  Noroxycodone(post dose2-4h) | 810.75 (419.08)
  Noroxycodone(post dose4-8h) | 1326.14 (645.18)
  Noroxycodone(post dose8-12h) | 1693.83 (978.49)
  Noroxycodone(post dose12-24h) | 2618.44 (1237.37)
  Hydroxymorphine(post dose0-2h) | 6.13 (8.11)
  Hydroxymorphine(post dose2-4h) | 30.16 (64.24)
  Hydroxymorphine(post dose4-8h) | 54.68 (67.67)
  Hydroxymorphine(post dose8-12h) | 72.85 (72.84)
  Hydroxymorphine(post dose12-24h) | 108.81 (77.11)
  Normethoxymorphone(post dose0-2h) | 130.63 (100.61)
  Normethoxymorphone(post dose2-4h) | 338.90 (241.50)
  Normethoxymorphone(post dose4-8h) | 601.46 (566.37)
  Normethoxymorphone(post dose8-12h) | 575.47 (287.77)
  Normethoxymorphone(post dose12-24h) | 796.81 (518.90)

ADVERSE EVENTS:
Time Frame: Single dose group the screening period is maximal 7 days, then 1 day dosing and sampling following by 1 day safety follow up, so total 9 days maximal. Multiple dose group the screening period is maximal 7 days, then 4 days dosing and sampleing following by 1 day safety follow up, so total 12 days maximal.
Description: No difference with the clinicaltrials.gov definition
Arm/Group | Oxycodone Hydrochloride Single Dose(5mg) | Oxycodone Hydrochloride Single Dose(10mg) | Oxycodone Hydrochloride Single Dose(20mg) | Oxycodone Hydrochloride Multiple Dose(10mg)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 8/15 | 11/15 | 14/15 | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Hydrochloride Single Dose(5mg) (N=15) | Oxycodone Hydrochloride Single Dose(10mg) (N=15) | Oxycodone Hydrochloride Single Dose(20mg) (N=15) | Oxycodone Hydrochloride Multiple Dose(10mg) (N=16)
Dizziness (Nervous system disorders) | 4 (4) | 10 (10) | 14 (14) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 10 (10) | 4 (4)
Drowsiness (Nervous system disorders) | 4 (4) | 3 (3) | 5 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 7 (7) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days